CLINICAL TRIAL: NCT00746564
Title: Confirm Implantable Cardiac Monitor Study
Brief Title: Study of New Implantable Loop Recorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 60020941D
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Tachyarrhythmias; Syncope
Keywords: Implantable Cardiac Monitor; Arrhythmias; Atrial Fibrillation
MeSH Terms: conditions — Tachycardia; Syncope; Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): SJM Confirm Device
  Interventions: Device: SJM Confirm

INTERVENTIONS:
Device: SJM Confirm — All patients in this study will receive the SJM Confirm device.

SUMMARY:
The goal of this IDE clinical study is to evaluate the quality of the cardiac signal recordings obtained by the St. Jude Medical (SJM) Confirm Implantable Cardiac Monitor (device).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have clinical syndromes or situations at increased risk of cardiac arrhythmias
* Patients who experience transient symptoms that may suggest a cardiac arrhythmia
* Patients who have been previously diagnosed with atrial fibrillation
* Patients who are suspected to have Atrial Fibrillation (AF) but AF has not been documented
* Patients who have provided written informed consent to participate in the study.

Exclusion Criteria:

* Patients who are under the age of 18 years
* Patients who have a life expectancy less than 1 year
* Patients who are unable to comply with the follow-up schedule
* Patients who are currently implanted with a pacemaker or defibrillator
* Patients who the physician deems inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Shipman, Study Director — Abbott Medical Devices
Locations (9):
- United States (9):
  - Alaska Heart Institute, Anchorage, Alaska
  - Arizona Arrhythmia Research, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - St. Jude Hospital, Fullerton, California
  - Scripps Clinic, La Jolla, California
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Providence- St Vincent Medical Center, Portland, Oregon
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- SJM Confirm Device: All patients in this study received the St. Jude Medical (SJM Confirm device.
Period: Overall Study
Arm/Group | SJM Confirm Device
Started | 75
Completed | 73
Not Completed | 2
Not completed — Required Pacemaker/ICD Implant | 2

BASELINE CHARACTERISTICS:
Population: All patients implanted with the Confirm Device.
Groups:
- Open Label: All patients who were implanted with the SJM Confirm device.
Arm/Group | Open Label
Number analyzed (Participants) | 75
Age, Continuous [Mean (Full Range); unit: years] | 62 [19 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity for R Waves During In-Clinic Recordings at Rest
Description: The sensitivity was calculated for each recording and for each subject.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I were included in this analysis. Total patients 48; 50-(1 withdrawal)-(1 patient with recording lacking the surface channel). Total analyzable recordings 88; 89-(1 recording lacking visible R waves).
Measure: Number (95% Confidence Interval); unit: percentage of recordings
Units Other Than Participants: Clinical recordings
Groups:
- SJM Confirm Device: All patients in this study received the SJM Confirm device.
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 48
Number analyzed (Clinical recordings) | 88
percentage of recordings | 100 [100 to 100]
Statistical Analysis 1: Comparison: SJM Confirm Device; The sensitivity was calculated for each recording and for each subject as follows: Amount of time (sec) R waves recorded on surface ECG were detected on in-clinic recordings/Total amount of time (sec) R waves were recorded on surface ECG; Test type: Superiority or Other; percentage of recordings = 100, 95% CI 2-sided [100 to 100]

2. Primary Outcome: Sensitivity for R Waves During In-Clinic Recordings During Treadmill Exercise
Description: The sensitivity for R waves during the in-clinic recordings was was calculated for each recording and for each subject.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 46; 50-(1 withdrawal)-(1 patient's recording lacking surface ECG channel)-(2 no recording obtained). Total analyzable recordings =39; 46 obtained-(7 with zero visible R waves).
Measure: Number (95% Confidence Interval); unit: percentage of recordings
Units Other Than Participants: Clinical Recordings
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 46
Number analyzed (Clinical Recordings) | 39
percentage of recordings | 98.1 [95.7 to 100]
Statistical Analysis 1: Comparison: SJM Confirm Device; The sensitivity was calculated for each recording during the treadmill test and for each subject as follows: Amount of time (sec) R waves recorded on surface ECG were detected on in-clinic recordings/Total amount of time (sec) R waves were recorded on surface ECG; Test type: Superiority or Other; percentage of clinical recordings = 98.1, 95% CI 2-sided [95.7 to 100]

3. Primary Outcome: Sensitivity for R Waves During In-Clinic Recordings During Hand to Hand/Shoulder Maneuvers
Description: The sensitivity for R waves during the in-clinic recordings was was calculated for each recording and for each subject.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 48; 50-(1 withdrawal)-(1 patient recording lacking surface ECG channel). Total analyzable recordings 82; 96 obtained-(14 recordings with zero visible R waves)=82 recordings
Measure: Number (95% Confidence Interval); unit: percentage of recordings
Units Other Than Participants: Clinical Recordings
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 48
Number analyzed (Clinical Recordings) | 82
percentage of recordings | 98.0 [95.5 to 100]
Statistical Analysis 1: Comparison: SJM Confirm Device; The sensitivity was calculated for each recording and for each subject during the hand to hand and hand to shoulder maneuvers as follows: Amount of time (sec) R waves recorded on surface ECG were detected on in-clinic recordings/Total amount of time (sec) R waves were recorded on surface ECG; Test type: Superiority or Other; percentage of recordings = 98.0, 95% CI 2-sided [95.5 to 100]

4. Primary Outcome: Positive Predictive Value (PPV) for In-Clinic Recordings at Rest
Description: The positive predictive value (PPV) for the in-clinic recording was calculated for each recording and for each subject.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 48; 50-(1 withdrawal)-(1 patient with no recording obtained). Total analyzable recordings 89.
Measure: Number (95% Confidence Interval); unit: percentage of recordings
Units Other Than Participants: Clinical Recordings
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 48
Number analyzed (Clinical Recordings) | 89
percentage of recordings | 98.9 [96.7 to 100]
Statistical Analysis 1: Comparison: SJM Confirm Device; The positive predictive value (PPV) was calculated for each recording and for each subject during the in-clinic recording at rest as follows: Amount of time (sec) R waves recorded on surface ECG were detected on in-clinic recording / Total amount of time (sec) R waves were recorded by device during in-clinic recording; Test type: Superiority or Other; percentage of recordings = 98.9, 95% CI 2-sided [96.7 to 100]

5. Primary Outcome: Positive Predictive Value (PPV) for In-Clinic Recordings During Treadmill Stress Test
Description: The positive predictive value (PPV) for the in-clinic recording was calculated for each recording and for each subject.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 45; 50-(1 withdrawal)-(1 patient recording lacking surface ECG channel)-(2 patients where no recording was obtained). Total analyzable recordings 45: 46 obtained-(1 recording with zero visible R waves).
Measure: Number (95% Confidence Interval); unit: percentage of recordings
Units Other Than Participants: Clinical recordings
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 45
Number analyzed (Clinical recordings) | 45
percentage of recordings | 77.1 [65.9 to 88.4]
Statistical Analysis 1: Comparison: SJM Confirm Device; The positive predictive value (PPV) was calculated for each recording and for each subject for the in-clinic recording during the treadmill exercise as follows: Amount of time (sec) R waves recorded on surface ECG were detected on in-clinic recording / Total amount of time (sec) R waves were recorded by device during in-clinic recording; Test type: Superiority or Other; percentage of recording = 77.1, 95% CI 2-sided [65.9 to 88.4]

6. Primary Outcome: Positive Predictive Value (PPV) During Hand to Hand/Shoulder Maneuvers
Description: The positive predictive value (PPV) for the in-clinic recording was was calculated for each recording and for each subject.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 48; 50-(1 withdrawal)-(1 patient recording lacking surface ECG channel). Total analyzable recordings 92: 96 obtained-(4 recordings with zero visible R waves)
Measure: Number (95% Confidence Interval); unit: percentage of recordings
Units Other Than Participants: Clinical Recordings
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 48
Number analyzed (Clinical Recordings) | 92
percentage of recordings | 85.0 [78.3 to 91.7]
Statistical Analysis 1: Comparison: SJM Confirm Device; The positive predictive value (PPV) was calculated for each recording and for each subject during Hand to Hand and Hand to Shoulder Maneuvers as follows: Amount of time (sec) R waves recorded on surface ECG were detected on in-clinic recording / Total amount of time (sec) R waves were recorded by device during in-clinic recording; Test type: Superiority or Other; Percentage of recordings = 85.0, 95% CI 2-sided [78.3 to 91.7]

7. Other Pre Specified Outcome: Interpretability of Weekly Subject Activator Recordings
Description: The proportion of recording time during which the device recording was interpretable was calculated for each weekly Patient Activator recording and for each subject. A random effects model was fitted to the data.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 30; 50-(1 withdrawal)-(19 patients who did not initiate recordings). Total analyzable recordings 58.
Measure: Number (95% Confidence Interval); unit: percentage of interpretable recordings
Units Other Than Participants: Clinical Recordings
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 30
Number analyzed (Clinical Recordings) | 58
percentage of interpretable recordings | 99.2 [98.5 to 100]
Statistical Analysis 1: Comparison: SJM Confirm Device; The proportion of recording time during which the device recording was interpretable was calculated for each weekly Patient Activator recording and for each subject as follows: Duration (sec) of interpretable recording / Total duration of recording time (sec); Test type: Superiority or Other; percentage of interpretable recording = 99.2, 95% CI 2-sided [98.5 to 100]

8. Other Pre Specified Outcome: Interpretability of Automatically Triggered/Symptom Driven Recordings
Description: The proportion of recording time during which the device recording was interpretable for each automatically triggered/symptom driven recording and for each subject.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 47; 50-(1 withdrawal)-(2 patients whose recordings were lost due to programming changes). Total analyzable recordings 2804.
Measure: Number (95% Confidence Interval); unit: percentage of interpretable recordings
Units Other Than Participants: Recordings
Groups:
- SJM Confirm Device: All patients implanted with an SJM Confirm device.
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 47
Number analyzed (Recordings) | 2804
percentage of interpretable recordings | 92.3 [91.9 to 92.6]
Statistical Analysis 1: Comparison: SJM Confirm Device; The proportion of recording time during which the device recording was interpretable for each automatically triggered/symptom driven recording and for each subject was calculated as follows: Duration of interpretable recording / Total duration of recording time; Test type: Superiority or Other; percentage of interpretable recording = 92.3, 95% CI 2-sided [91.9 to 92.6]

9. Other Pre Specified Outcome: Inappropriateness of Automatically Triggered Recordings - Phase I
Description: The proportion of automatically triggered recordings that were inappropriate (i.e. noise triggered)was calculated and reported using a generalized estimating equation (GEE) model for binomial outcomes to account for multiple recordings per patient.
Time Frame: 6 weeks
Population: 50 patients implanted with the SJM Confirm device in Phase I. Total patients 47; 50-(1 withdrawal)-(2 patients whose recordings were lost due to programming changes).
Measure: Number (95% Confidence Interval); unit: percentage of inappropriate recordings
Units Other Than Participants: Recordings
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 47
Number analyzed (Recordings) | 2741
percentage of inappropriate recordings | 86.2 [79.4 to 91.0]
Statistical Analysis 1: Comparison: SJM Confirm Device; Test type: Superiority or Other; percentage of inappropriate recordings = 86.2, 95% CI 2-sided [79.4 to 91.0]

10. Other Pre Specified Outcome: Inappropriateness of Automatically Triggered Recordings - Phase II
Description: The proportion of automatically triggered recordings that were inappropriate (i.e. noise triggered)was calculated and reported using a GEE model for binomial outcomes to account for multiple recordings per patient.
Time Frame: 6 weeks
Population: All patients implanted with the SJM Confirm device in participating in Phase II. Total patients 36: (19 rollovers from Phase I enrollments)+(25 Phase II enrollments)-(1 withdrawal)-(7 subjects with no automatically triggered recordings). Total recordings obtained: 958
Measure: Number (95% Confidence Interval); unit: percentage of inappropriate recordings
Units Other Than Participants: Recording
Groups:
- SJM Confirm Device: All patients implanted with the SJM Confirm device.
Arm/Group | SJM Confirm Device
Number analyzed (Participants) | 36
Number analyzed (Recording) | 958
percentage of inappropriate recordings | 62.3 [48.1 to 76.2]
Statistical Analysis 1: Comparison: SJM Confirm Device; Test type: Superiority or Other; percentage of inappropriate recordings = 63.2, 95% CI 2-sided [48.1 to 76.2]

ADVERSE EVENTS:
Time Frame: Baseline, 6-Week, 3-Month, and every 6 Months for the duration of the study or up to 5 years.
Description: Patients were assessed for adverse events, and the Confirm device was evaluated at each study visit.
Arm/Group | SJM Confirm Device
Serious Adverse Events (participants affected / at risk) | 11/75
Other Adverse Events (participants affected / at risk) | 14/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJM Confirm Device (N=75)
PREMATURE BATTERY DEPLETION/ ICM (Surgical and medical procedures) | 10 (10)
DEVICE EXTRUSION (Surgical and medical procedures) | 1 (1)
VAGAL REACTION (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJM Confirm Device (N=75)
EARLY BATTERY DEPLETION/ PATIENT ACTIVATOR (Surgical and medical procedures) | 4 (4)
Excessive Noise on the EGM Resulting in Inability to Interpret the EGM (Surgical and medical procedures) | 7 (12)
Undersensing (Surgical and medical procedures) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less